CLINICAL TRIAL: NCT01084863
Title: A Double-Blind, Randomized, Parallel Phase I/IIb Study to Evaluate Initial Safety and Efficacy, Comparative Pharmacokinetics, and Immunogenicity for CT-P6 and Herceptin in Metastatic Breast Cancer
Brief Title: Evaluate Safety, Efficacy and Pharmacokinetics
Acronym: Compare
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CT-P6/1.1
Record Dates: First submitted 2010-03-05; First posted 2010-03-11 (Estimated); Results first posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Breast Cancer
Keywords: Herceptin; Her 2-positive; metastatic breast cancer; CT-P6
MeSH Terms: conditions — Breast Neoplasms | interventions — CT-P6; Trastuzumab; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CT-P6 & Paclitaxel (Experimental): CT-P6 was administered at a loading dose of 8 mg/kg body weight by IV infusion over 90 minutes on Day 1, Cycle 1, then at 6 mg/kg repeated at 3-weekly intervals until disease progression, death, or discontinuation.
  Paclitaxel was administered at a dose of 175 mg/m2 body surface area (BSA) as a continuous 3-hour IV infusion on the day following the first dose of study drug (CT-P6). If the first dose of study drug was well tolerated, subsequent doses of paclitaxel were given immediately after the next dose of study drug. Paclitaxel cycles were repeated every 3 weeks until disease progression, death, intolerable toxicity, or discontinuation.
  Interventions: Drug: CT-P6; Drug: Paclitaxel
- Herceptin & Paclitaxel (Active Comparator): Herceptin was administered at a loading dose of 8 mg/kg body weight by IV infusion over 90 minutes on Day 1, Cycle 1, then at 6 mg/kg repeated at 3-weekly intervals until disease progression, death, or discontinuation.
  Paclitaxel was administered at a dose of 175 mg/m2 body surface area (BSA) as a continuous 3-hour IV infusion on the day following the first dose of study drug (Herceptin). If the first dose of study drug was well tolerated, subsequent doses of paclitaxel were given immediately after the next dose of study drug. Paclitaxel cycles were repeated every 3 weeks until disease progression, death, intolerable toxicity, or discontinuation.
  Interventions: Drug: Herceptin; Drug: Paclitaxel

INTERVENTIONS:
Drug: CT-P6 — CT-P6: administered every 3 weeks
  Arms: CT-P6 & Paclitaxel
Drug: Herceptin — Herceptin: administered every 3 weeks
  Other Names: Trastuzumab
  Arms: Herceptin & Paclitaxel
Drug: Paclitaxel — Paclitaxel: administered every 3 weeks

SUMMARY:
The purpose of the study is to demonstrate equivalent pharmacokinetics (PK)

DETAILED DESCRIPTION:
Patients will receive CT-P6 or Herceptin.

ELIGIBILITY:
Inclusion Criteria:

* Are females
* Have a Her 2 over-expression
* Have Eastern Cooperative Oncology Group (ECOG) 0 or 1

Exclusion Criteria:

* Current clinical or radiographic evidence central nervous system (CNS) metastases
* Current Known infection
* Pregnant or nursing mother

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2023-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Investigational Site, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Period: Main Study Treatment Period
Arm/Group | CT-P6 & Paclitaxel | Herceptin & Paclitaxel
Started | 76 | 67
Completed | 60 | 56
Not Completed | 16 | 11
Not completed — Disease progression | 11 | 7
Not completed — Adverse Event | 5 | 3
Not completed — Other Reason | 0 | 1
Period: Treatment Period Beyond Cycle 8
Arm/Group | CT-P6 & Paclitaxel | Herceptin & Paclitaxel
Started (Of these, 7 patients who completed Main Study Treatment Period (Cycle 8) but discontinued treatment before Cycle 9 were also counted in the Treatment Period Beyond Cycle 8.) | 60 | 56
Completed | 0 | 0
Not Completed | 60 | 56
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Physician Decision | 2 | 4
Not completed — Disease progression | 51 | 45
Not completed — Adverse Event | 1 | 0
Not completed — Other | 0 | 1
Not completed — Other reason | 2 | 2

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) was defined as all randomized patients who received any study drug (CT-P6 or Herceptin) and had at least one post-baseline assessment, with the exception of the patients who violated against Herceptin indication.
Groups:
- CT-P6 & Paclitaxel: CT-P6 was administered at a loading dose of 8 mg/kg body weight by IV infusion over 90 minutes on Day 1, Cycle 1, then at 6 mg/kg repeated at 3-weekly intervals until disease progression, death, or discontinuation.
  Paclitaxel was administered at a dose of 175 mg/m2 BSA as a continuous 3-hour IV infusion on the day following the first dose of study drug (CT-P6). If the first dose of study drug was well tolerated, subsequent doses of paclitaxel were given immediately after the next dose of study drug. Paclitaxel cycles were repeated every 3 weeks until disease progression, death, intolerable toxicity, or discontinuation.
- Herceptin & Paclitaxel: Herceptin was administered at a loading dose of 8 mg/kg body weight by IV infusion over 90 minutes on Day 1, Cycle 1, then at 6 mg/kg repeated at 3-weekly intervals until disease progression, death, or discontinuation.
  Paclitaxel was administered at a dose of 175 mg/m2 BSA as a continuous 3-hour IV infusion on the day following the first dose of study drug (Herceptin). If the first dose of study drug was well tolerated, subsequent doses of paclitaxel were given immediately after the next dose of study drug. Paclitaxel cycles were repeated every 3 weeks until disease progression, death, intolerable toxicity, or discontinuation.
- Total: Total of all reporting groups
Arm/Group | CT-P6 & Paclitaxel | Herceptin & Paclitaxel | Total
Number analyzed (Participants) | 76 | 67 | 143
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 63 | 59 | 122
  >=65 years | 13 | 8 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (10.26) | 53.6 (10.47) | 54.4 (10.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 67 | 143
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 45 | 35 | 80
  Asian | 31 | 32 | 63
Region of Enrollment [Count of Participants; unit: Participants]
  Bulgaria | 6 | 2 | 8
  South Korea | 31 | 32 | 63
  Latvia | 7 | 6 | 13
  Russia | 19 | 16 | 35
  Serbia | 4 | 5 | 9
  Ukraine | 9 | 6 | 15
Childbearing potential [Count of Participants; unit: Participants]
  Yes | 18 | 24 | 42
  No | 58 | 43 | 101
Height at Screening [Mean (Standard Deviation); unit: cm] | 158.9 (6.70) | 160.3 (7.20) | 159.6 (6.95)
Weight at Screening [Mean (Standard Deviation); unit: kg] | 66.0 (16.64) | 67.6 (15.71) | 66.7 (16.17)
BSA at Screening [Mean (Standard Deviation); unit: m2] | 1.70 (0.22) | 1.73 (0.22) | 1.71 (0.22)
Prior chemotherapy [Count of Participants; unit: Participants]
  Yes | 29 | 26 | 55
  No | 47 | 41 | 88
Eastern Cooperative Oncology Group (ECOG) performance status [Count of Participants; unit: Participants] — ECOG performance status was performed based on the values collected for randomization. All patients had a grade 0 or 1 ECOG performance based on the values collected for randomization. Grade 0 (Fully active, able to carry on all pre-disease performance without restriction), Grade 1 (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work)
  Participants
    0 | 35 | 25 | 60
    1 | 41 | 42 | 83
Karnofsky performance status [Count of Participants; unit: Participants] — Karnofsky performance status was performed based on the values collected for randomization. Category 1 (80-100 points) = Able to carry on normal activity and to work; no special care needed, Category 2 (50-70 points) = Unable to work; able to live at home and care for most personal needs; varying amount of assistance needed, Category 3 (0-40 points) = Unable to care for self; requires equivalent of institutional or hospital care; disease may be progressing rapidly.
  Participants
    Category 1 | 72 | 62 | 134
    Category 2 | 1 | 3 | 4
    Category 3 | 0 | 0 | 0
    Not reported | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration Time Curve at Steady State (AUCss)
Description: Area under the concentration time curve at steady state (AUCss), defined as area under the concentration-time curve between Cycle 8 to Cycle 9. The primary endpoint was reached at 6 months (8 treatment cycle; Main Study Treatment Period).
Time Frame: 3, 6, 12, 24, 72, 168, 336, 504 hours predose
Population: PK Analysis Set - Global (PKASg) was defined as all FAS patients who had achieved steady state by the 8th cycle, which required three consecutive similar trough concentrations.
Measure: Mean (Standard Deviation); unit: ug*h/mL
Arm/Group | CT-P6 & Paclitaxel | Herceptin & Paclitaxel
Number analyzed (Participants) | 51 | 49
ug*h/mL | 34400 (15000) | 31800 (9820)
Statistical Analysis 1: Comparison: CT-P6 & Paclitaxel vs Herceptin & Paclitaxel; Test type: Equivalence — Pharmacokinetic equivalence was predefined based on acceptance criteria, 80% to 125%; Geometric Mean Ratio = 104.57, 90% CI 2-sided [93.64 to 116.78]

2. Secondary Outcome: Trough Concentration at Steady State (CtroughSS)
Description: Trough concentration at steady state (CtroughSS), defined as trough concentration at steady state. The secondary endpoint was reached at 6 months (8 treatment cycle; Main Study Treatment Period).
Time Frame: 3, 6, 12, 24, 72, 168, 336, 504 hours predose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | CT-P6 & Paclitaxel | Herceptin & Paclitaxel
Number analyzed (Participants) | 51 | 49
ug/mL | 21.1 (7.83) | 20.8 (8.26)

3. Secondary Outcome: Cardiotoxicity
Description: Cardiac Ejection Fraction Assessment, defined as Mean change from baseline to endpoint assessment in left ventricular ejection fraction (LVEF, Unit: %) from the independent tumor review committee (ITRC).
Time Frame: Up to approximately 1 year
Population: Safety Analysis Set (SAF) was defined as all patients in the FAS. All patients receiving at least one dose of CT-P6 were analyzed under the CT-P6 treatment group. All other patients were analyzed under the Herceptin treatment group.
Measure: Mean (Standard Deviation); unit: %; percentage of LVEF
Arm/Group | CT-P6 & Paclitaxel | Herceptin & Paclitaxel
Number analyzed (Participants) | 62 | 53
%; percentage of LVEF | -5.49 (6.543) | -6.43 (5.622)

4. Secondary Outcome: Immunogenicity
Description: Immunogenicity, defined as proportion of patients with antibodies to study drug (positive for antidrug antibody [ADA] result after the first study infusion).
Time Frame: every 4 cycles (each cycle is 3 weeks), Up to approximately 5.5 years
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P6 & Paclitaxel | Herceptin & Paclitaxel
Number analyzed (Participants) | 76 | 67
Participants | 2 | 0

5. Secondary Outcome: Overall Response Rate (ORR; Complete Response [CR] Plus Partial Response [PR]) as Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: Overall response rate (ORR) based on best overall response (BOR) during the Main Study Treatment Period and up to 1-year treatment from the independent tumor review committee (ITRC) and Investigator.
  ORR (complete response [CR] plus partial response [PR]), as assessed by Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1 To be assigned a best ORR of PR or CR, changes in tumour assessments must be confirmed no less than 4 weeks after the criteria for response were met.
Time Frame: every 6 weeks (up to cycle 4) or 12 weeks (after cycle 4) (every cycle is 3 weeks), up to 6 months in Main treatment period and up to 1 year
Population: Full Analysis Set (FAS) was defined as all randomized patients who received any study drug (CT-P6 or Herceptin) and had at least one post-baseline assessment, with the exception of the patients who violated against Herceptin indication.
Measure: Number; unit: percentage of responder
Groups:
- CT-P6 & Paclitaxel ITRC; CT-P6 & Paclitaxel Investigator: CT-P6 was administered at a loading dose of 8 mg/kg body weight by IV infusion over 90 minutes on Day 1, Cycle 1, then at 6 mg/kg repeated at 3-weekly intervals until disease progression, death, or discontinuation.
  Paclitaxel was administered at a dose of 175 mg/m2 BSA as a continuous 3-hour IV infusion on the day following the first dose of study drug (CT-P6). If the first dose of study drug was well tolerated, subsequent doses of paclitaxel were given immediately after the next dose of study drug. Paclitaxel cycles were repeated every 3 weeks until disease progression, death, intolerable toxicity, or discontinuation.
- Herceptin & Paclitaxel ITRC; Herceptin & Paclitaxel Investigator: Herceptin was administered at a loading dose of 8 mg/kg body weight by IV infusion over 90 minutes on Day 1, Cycle 1, then at 6 mg/kg repeated at 3-weekly intervals until disease progression, death, or discontinuation.
  Paclitaxel was administered at a dose of 175 mg/m2 BSA as a continuous 3-hour IV infusion on the day following the first dose of study drug (Herceptin). If the first dose of study drug was well tolerated, subsequent doses of paclitaxel were given immediately after the next dose of study drug. Paclitaxel cycles were repeated every 3 weeks until disease progression, death, intolerable toxicity, or discontinuation.
Arm/Group | CT-P6 & Paclitaxel ITRC | Herceptin & Paclitaxel ITRC | CT-P6 & Paclitaxel Investigator | Herceptin & Paclitaxel Investigator
Number analyzed (Participants) | 76 | 67 | 76 | 67
percentage of responder
  Main Study Treatment Period | 61.8 | 76.1 | 68.4 | 80.6
  1 Year | 65.8 | 77.6 | 72.4 | 80.6

6. Secondary Outcome: Serum Human Epidermal Growth Factor Receptor-2 (HER-2) Shed Antigen Value
Description: Serum Human epidermal growth factor receptor-2 (HER-2) shed antigen values at baseline (Cycle 1, Day 1) and the last assessments.
Time Frame: day 1 of each cycle (every cycle is 3 weeks), Up to approximately 5.5 years
Population: Safety Analysis Set (SAF) was defined as all patients in the FAS. All patients receiving at least one dose of CT-P6 were analyzed under the CT-P6 treatment group. All other patients were analyzed under the Herceptin treatment group.
  One subject in the CT-P6 treatment group did not have baseline HER-2 Shed antigen result.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CT-P6 & Paclitaxel | Herceptin & Paclitaxel
Number analyzed (Participants) | 76 | 67
ng/mL
  Baseline (Cycle 1, Day 1): number analyzed (Participants) | 75 | 67
  Baseline (Cycle 1, Day 1) | 85.20 (195.10) | 77.87 (169.14)
  Last assessment | 49.68 (162.10) | 8.82 (19.97)

ADVERSE EVENTS:
Time Frame: Adverse event (AE) reporting extended from the date of informed consent until completion of the final visit. (Up to approximately 170 months)
Arm/Group | CT-P6 & Paclitaxel | Herceptin & Paclitaxel
All-Cause Mortality (participants affected / at risk) | 2/76 | 3/67
Serious Adverse Events (participants affected / at risk) | 12/76 | 19/67
Other Adverse Events (participants affected / at risk) | 74/76 | 64/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CT-P6 & Paclitaxel (N=76) | Herceptin & Paclitaxel (N=67)
Acute tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 2 (2) | 0 (0)
Biliary drainage (Surgical and medical procedures) | 0 (0) | 1 (4)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (3)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 1 (1) | 5 (5)
Endoscopic retrograde cholangiopancreatography (Investigations) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Hepatitis cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Neutropenic infection (Infections and infestations) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (2)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CT-P6 & Paclitaxel (N=76) | Herceptin & Paclitaxel (N=67)
Abdominal pain (Gastrointestinal disorders) | 4 (7) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 8 (13)
Alanine aminotransferase increased (Investigations) | 7 (12) | 8 (19)
Alopecia (Skin and subcutaneous tissue disorders) | 47 (59) | 44 (50)
Anaemia (Blood and lymphatic system disorders) | 9 (19) | 5 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (33) | 15 (29)
Aspartate aminotransferase increased (Investigations) | 6 (8) | 7 (16)
Asthenia (General disorders) | 24 (52) | 10 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (7) | 11 (19)
Blood alkaline phosphatase increased (Investigations) | 5 (9) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 13 (22) | 6 (10)
Breast pain (Reproductive system and breast disorders) | 4 (5) | 2 (2)
Chills (General disorders) | 6 (11) | 7 (8)
Constipation (Gastrointestinal disorders) | 4 (6) | 10 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 8 (11)
Decreased appetite (Metabolism and nutrition disorders) | 7 (12) | 8 (22)
Diarrhoea (Gastrointestinal disorders) | 13 (23) | 18 (38)
Dizziness (Nervous system disorders) | 6 (11) | 13 (23)
Dyspepsia (Gastrointestinal disorders) | 5 (6) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 5 (7)
Face oedema (General disorders) | 2 (3) | 4 (5)
Fatigue (General disorders) | 10 (27) | 10 (31)
Gamma-glutamyltransferase increased (Investigations) | 5 (13) | 2 (6)
Headache (Nervous system disorders) | 11 (16) | 13 (18)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (13) | 3 (13)
Hypertension (Vascular disorders) | 5 (6) | 4 (9)
Insomnia (Psychiatric disorders) | 7 (14) | 13 (16)
Left ventricular dysfunction (Cardiac disorders) | 2 (2) | 5 (7)
Leukopenia (Blood and lymphatic system disorders) | 8 (10) | 12 (28)
Mucosal inflammation (General disorders) | 4 (5) | 5 (6)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 7 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 31 (134) | 31 (127)
Nail disorder (Skin and subcutaneous tissue disorders) | 2 (3) | 4 (4)
Nasopharyngitis (Infections and infestations) | 7 (11) | 3 (9)
Nausea (Gastrointestinal disorders) | 19 (51) | 17 (41)
Neuropathy peripheral (Nervous system disorders) | 23 (46) | 21 (54)
Neutropenia (Blood and lymphatic system disorders) | 32 (59) | 33 (85)
Oedema peripheral (General disorders) | 8 (10) | 8 (12)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 5 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (14) | 17 (32)
Paraesthesia (Nervous system disorders) | 4 (4) | 2 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 21 (79) | 27 (50)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (11) | 12 (18)
Pyrexia (General disorders) | 10 (18) | 10 (18)
Rash (Skin and subcutaneous tissue disorders) | 10 (16) | 12 (29)
Stomatitis (Gastrointestinal disorders) | 6 (13) | 11 (14)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 6 (10)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (7)
Vomiting (Gastrointestinal disorders) | 5 (10) | 9 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes